CLINICAL TRIAL: NCT01467089
Title: The Assessment of Movement Disorders Utilizing Live Two-Way Video
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Sandeep kapoor, Principal Investigator, Northwell Health
Other Study IDs: 11-243B
Record Dates: First submitted 2011-10-31; First posted 2011-11-08 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Tardive Dyskinesia
Keywords: Schizophrenia; Extrapyramidal symptoms; Tardive dyskinesia; Two Way Video Assessment
MeSH Terms: conditions — Tardive Dyskinesia; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- schizophrenia: Inclusion Criteria: Inpatients and outpatients aged 18-75 years old who have been taking antipsychotics for longer than 6 months in their life time, and that have been compliant for the past week. Patients will be referred by their treating doctors if they have some evidence of movement disorder based on the physician's clinical judgment. We will also include 25% of the sample without any evidence of movement disorder.
  Exclusion Criteria: Patients who have medical conditions which make it difficult to perform a physical examination. Patients who are clinically too ill to consent and/or unable to cooperate with the examination procedures.
  Interventions: Other: Two way video assessment

INTERVENTIONS:
Other: Two way video assessment — Participants will be assessed extrapyramidal symptoms and tardive dyskinesia

SUMMARY:
The purpose of this project is to determine the equivalency of extrapyramidal symptoms (EPS) and tardive dyskinesia (TD) examinations conducted via live two-way video versus live examinations completed in-person

DETAILED DESCRIPTION:
Extrapyramidal symptoms (EPS) and tardive dyskinesia (TD) are one of the most frequent and troublesome adverse events when taking antipsychotic agents. The investigators aim in this study to determine if the investigators can conduct examinations for EPS and TD remotely using live two-way video. It is potentially beneficial for patients, especially those who are located far away from psychiatrists if they could be seen by trained clinicians and assessed for EPS and TD via two-way video in the future. Participants will be asked to have a medical assessment which consists of simple questions and some examination of their movements via two-way video and in person. The investigators will compare the results of video examinations with the results of live examinations.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients aged 18-75 years old who have been taking antipsychotics for longer than 6 months in their life time, and
* That have been compliant for the past week.

Exclusion Criteria:

* Patients who have medical conditions which make it difficult to perform a physical examination.
* Patients who are clinically too ill to consent and/or unable to cooperate with the examination procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients with schizophrenia will be recruited via in- and outpatient psychiatry service of The Zucker Hillside Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Abnormal Involuntary Movement Scale (AIMS) when done in-person versus via two-way video | Baseline
Modified Simpson Angus Scale (mSAS) short version when done in-person versus via two-way video | Baseline

SECONDARY OUTCOMES:
the correlation between the short version and full version of the Modified Simpson Angus Scale (mSAS) | Baseline
  total score of short version-Modified Simpson Angus Scale vs. total score of full version-Modified Simpson Angus Scale

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Kapoor, MD, Principal Investigator — Northwell Health
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States